CLINICAL TRIAL: NCT01116076
Title: DECISION+: Une Formation Pour Les médecins de Famille Sur la Prise de décision partagée Afin d'Optimiser Les décisions Cliniques Concernant l'Utilisation d'Antibiotiques Pour Les Infections aiguës Des Voies Respiratoires (IAVR)
Brief Title: DECISION+, a Training Program to Improve Optimal Drug Prescription
Acronym: Decision+
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: CHU de Quebec-Universite Laval (Other)
Responsible Party: Principal Investigator, France Legare, Canada Research Chair in Implementation of Shared Decision Making in Primary Care, CHU de Quebec-Universite Laval
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: FRSQ20131; 35247 (Other: CHUQ)
Record Dates: First submitted 2010-05-03; First posted 2010-05-04 (Estimated); Last update posted 2013-02-01 (Estimated); Status verified 2013-01

CONDITIONS: Acute Respiratory Infections

ARMS (2):
- DECISION+ Program (Experimental): Exposure to the Decision+ Program
  Interventions: Behavioral: Decision+ program (to improve optimal drug prescription for ARI)
- Control (No Intervention): Usual Care

INTERVENTIONS:
Behavioral: Decision+ program (to improve optimal drug prescription for ARI) — DECISION+ is a multifaceted intervention program that includes: On site course and Internet-based courses (2x120 min), reminders of expected behaviours and feedback.
  Arms: DECISION+ Program

SUMMARY:
Decisions about the use of antibiotics for acute respiratory infections are the most frequently reported reason for consulting a family physician. Although it varies according to the specific type of acute respiratory infections, the use of antibiotics is estimated to be 63% to 67%, well above the expected prevalence of bacterial infections thus suggesting overuse of antibiotics. Consequently, there is an urgent need for helping family physicians and their patients to improve the clinical decision making process regarding the use of antibiotics for acute respiratory infections. We will evaluate the impact of DECISION +, a multifaceted intervention program that includes training in shared decision making, reminders and feedback targeting physicians, and decision support tools targeting patients on the decision to use antibiotics for acute respiratory infections. Results from this study will lay the ground for a national strategy targeting the improvement of the clinical decision making process regarding antibiotic use for acute respiratory infections in primary care. In turn, this will increase quality of care and patient safety.

ELIGIBILITY:
FAMILY PHYSICIANS:

Inclusion Criteria:

* All FP (teachers and residents) providing care in the walk-in clinic in each Family Practice Teaching Unit (FPTU) will be eligible to participate in the trial.

Exclusion Criteria:

* he/she was involved or participated in the DECISION + pilot RCT
* he/she is not expected to be practicing at the FPTU for the whole duration of the study (e.g. residents ending their residency program or doing rotations outside of the FPTU, planned pregnancy/delivery, planned retirement).

PATIENTS:

Inclusion Criteria:

* if 17 years old and under, must be accompanied by a parents or a guardians)
* they are consulting a participating physician for an ARI, for which treatment with an antibiotic is considered
* they are able (patients or the accompanying parent or guardians) to read, understand and write French (expected level: 8th grade)
* they give informed consent

Exclusion Criteria:

* Patients with a condition requiring emergency care will be excluded.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 712 (Actual)
Dates: Start 2010-05; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
Proportion of patients reporting a decision for "immediate antibiotics." | After index consultation

SECONDARY OUTCOMES:
Decision to use antibiotics | After index consultation
  After an index consultation, we will ask patients: "Was a prescription for an antibiotic or a sample of antibiotic provided to treat an ARI (acute otitis media, acute bronchitis, acute pharyngitis, or acute rhinosinusitis)?" Possible answers will be:
  * Yes,(Immediate antibiotics);
  * Yes,(Delayed antibiotics);
  * No (no antibiotics).
Decisional conflict | After index consultation
  Will be assessed with the Decisional Conflict Scale (DCS) after the index consultation. This questionnaire is similar for physicians and patients and includes 19 items, on a five-point Likert scale, divided into five subscales that are i)uncertainty and its modifiable deficits: ii) knowledge, iii) values clarification, iv) support and v) perception of an effective choice. Both the physician and patient versions of the DCS have adequate psychometric properties and have the same meaning for both physicians and patients.
Adherence to the decision that was made | 2 weeks after the index consultation
  2 weeks after the index consultation, patients will be asked via a telephone interview: "What was the decision made with the FP about antibiotic use for ARI two weeks ago?" and "Have you complied with this decision?" (yes or no). If patients answer "no", research assistants, using an open-ended question, will inquire about the reasons and the options that were adhered to. Interviewers will be unaware of the study group and will be instructed not to ask questions that could reveal the study group.
Decisional regret | 2 weeks after the index consultation
  2 weeks after the index consultation, decisional regret will be assessed in patients using the Decisional Regret Scale (DRS) via a telephone interview. The DRS is a 5-item scale with adequate psychometric properties that correlates strongly with decision satisfaction and overall QOL.
Quality of life (QOL) | Baseline and 2 weeks after the index consultation
  For patients only, before and two weeks after the index consultation (via a telephone interview), QOL will be assessed using the Short Form-12 (SF-12V2 Health survey). This questionnaire measures general health status from the patient's point of view and includes eight concepts commonly represented in health status: physical functioning, role functioning, bodily pain, general health, vitality, social functioning, and emotional and mental health.
Intention to engage in SDM in future consultations dealing with antibiotic use for ARI | Baseline and 2 weeks after the index consultation
  In FP and their patients, this intention will be assessed based on the Theory of planned behavior (TPB). The questionnaire includes 15 items, on a 7-point Likert scale, that cover the constructs of the TPB, namely attitudes, social norm, perceived behavioral control and intention. Patients will complete this questionnaire before and 2 weeks after the index consultation; physicians will complete it once during the baseline data collection period and after the last encounter of the post-intervention data collection period.

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier Université Laval - Hôpital St-François d'Assise, Québec, Quebec, Canada

REFERENCES:
- [Background] Legare F, Labrecque M, Godin G, LeBlanc A, Laurier C, Grimshaw J, Castel J, Tremblay I, Fremont P, Cauchon M, Lemieux K, Rheaume C. Training family physicians and residents in family medicine in shared decision making to improve clinical decisions regarding the use of antibiotics for acute respiratory infections: protocol for a clustered randomized controlled trial. BMC Fam Pract. 2011 Jan 26;12:3. doi: 10.1186/1471-2296-12-3. PMID 21269509
- [Result] Legare F, Labrecque M, Cauchon M, Castel J, Turcotte S, Grimshaw J. Training family physicians in shared decision-making to reduce the overuse of antibiotics in acute respiratory infections: a cluster randomized trial. CMAJ. 2012 Sep 18;184(13):E726-34. doi: 10.1503/cmaj.120568. Epub 2012 Jul 30. PMID 22847969
- [Derived] Legare F, Guerrier M, Nadeau C, Rheaume C, Turcotte S, Labrecque M. Impact of DECISION + 2 on patient and physician assessment of shared decision making implementation in the context of antibiotics use for acute respiratory infections. Implement Sci. 2013 Dec 26;8:144. doi: 10.1186/1748-5908-8-144. PMID 24369771
- [Derived] Guerrier M, Legare F, Turcotte S, Labrecque M, Rivest LP. Shared decision making does not influence physicians against clinical practice guidelines. PLoS One. 2013 Apr 24;8(4):e62537. doi: 10.1371/journal.pone.0062537. Print 2013. PMID 23638111
- See also: Related Info — http://decision.chaire.fmed.ulaval.ca/index.php?id=66&L=2